CLINICAL TRIAL: NCT05979597
Title: The Effect of Adjuvant Dexamethasone on Postoperative Pain, Analgesic Consumption and Block Properties in Suprainguinal Fascia Iliaca Block (SFIB) in Knee Arthroplasty
Brief Title: The Effect of Adjuvant Dexamethasone on Postoperative Pain, Analgesic Consumption and Block Properties in SFIB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsun Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Hale Kefeli Celik, Anesthesiologist, Principal Investigator, Samsun Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SFIB-TEZ
Record Dates: First submitted 2023-07-29; First posted 2023-08-07 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Regional Anesthesia
Keywords: regional anesthesia; suprainguinal fascia iliaca block; dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The patient will not know which study group he is in. The anesthetist, who will perform the regional block, will give the block to be applied in a sealed envelope by an assistant staff outside the study, and at the same time, the patient will not know which block has been made. The anesthesiologist who made the block will not participate in the pain follow-up of the patients. Postoperative pain assessment and data collection will be performed by another investigator blinded to the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group SFIB (Suprainguinal fascia iliaca block) (Active Comparator): In the patient lying in the supine position, a high-frequency linear probe is inserted under sterile conditions, using an in-plane technique, 1 cm cephalad of the inguinal ligament with a needle. Using hydro-dissection, the fascia iliaca is separated from the iliac muscle and a space is created where the needle can be advanced cranially, and the procedure will be completed by injecting local anesthetic into this space.
  Interventions: Procedure: Suprainguinal fascia iliaca block
- Group SFIB+dexa (Suprainguinal fascia iliaca block+dexamethasone) (Active Comparator): In the patient lying in the supine position, a high-frequency linear probe is inserted under sterile conditions, using an in-plane technique, 1 cm cephalad of the inguinal ligament with a needle. Using hydro-dissection, the fascia iliaca is separated from the iliac muscle and a space is created where the needle can be advanced cranially, and the procedure will be completed by injecting local anesthetic+dexamethasone into this space.
  Interventions: Procedure: Suprainguinal fascia iliaca block+dexamethasone

INTERVENTIONS:
Procedure: Suprainguinal fascia iliaca block — After the operation is completed, the fascia iliaca will be separated from the iliacus muscle. With ultrasound guidance, the local anesthetic injection will be made between the fascia and the muscle.
  Arms: Group SFIB (Suprainguinal fascia iliaca block)
Procedure: Suprainguinal fascia iliaca block+dexamethasone — After the operation is completed, the fascia iliaca will be separated from the iliacus muscle. With ultrasound guidance, the local anesthetic+dexamethasone injection will be made between the fascia and the muscle.
  Arms: Group SFIB+dexa (Suprainguinal fascia iliaca block+dexamethasone)

SUMMARY:
The investigators aimed to demonstrate that dexamethasone added as an adjuvant to local anaesthetic agent in suprainguinal fascia iliaca block for effective postoperative analgesia after knee arthroplasty would prolong the duration of sensory block and reduce postoperative pain intensity and analgesic consumption.

DETAILED DESCRIPTION:
Total knee arthroplasty is one of the major orthopedic surgeries that cause severe postoperative pain. A successful post-operative outcome is possible with strong and effective pain control followed by early mobilization and a good functional recovery. Suprainguinal fascia iliaca plan block (SFIB) has been shown to be an effective postoperative method in multimodal analgesia regime in lower extremity surgery. It has been reported in the literature that dexamethasone added to local anaesthetics in peripheral nerve blocks prolongs the duration of sensory block, improves the quality of analgesia, reduces postoperative pain intensity and opioid consumption.

In this study, the investigators aimed to demonstrate that dexamethasone added as an adjuvant to local anaesthetic agent in SFIB for effective postoperative analgesia after knee arthroplasty would prolong the duration of sensory block and reduce postoperative pain intensity and analgesic consumption.

An identification number will be randomly assigned to each participants, whose written consent was obtained before the surgery, when they are admitted to the postoperative recovery room. In the postoperative period, participants will be followed up with these numbers. Which group the participants will be included in will be determined by the closed envelope method.

Participants undergoing unilateral knee arthroplasty will be included in the study. Following the end of surgery, the participants will be divided into two groups in the recovery room and SFIB will be applied to both groups. Participants in group SFIB will receive 0.25% bupivacaine as local anaesthetic. Participants in group SFIB+dexamethasone will receive 0.25% bupivacaine as local anaesthetic and 8 mg dexamethasone as adjuvant.

The participant with the block will be followed in the recovery room and if the block is successful, morphine patient controlled analgesia (PCA) treatment will be started and the participant will be taken to the ward. A standard analgesia regimen (1 g iv paracetamol every 8 hours, 50 mg iv dexketoprofen every 12 hours) was used in all participants.

Evaluation of postoperative pain will be done with numerical rating scale (NRS). Pain levels will be questioned in two different ways as rest and passive moving.

ELIGIBILITY:
Inclusion Criteria:

* Having undergone unilateral knee replacement surgery under elective conditions,
* Age range of 18-75 years,
* American Society of Anesthesiologist's physiologic state I-III patients,
* written consent who agreed to participate in the study.

Exclusion Criteria:

* BMI>35
* who do not want to be included in the study by not signing the voluntary consent form,
* Local infection, hematoma, hernia, neoplasm etc. in the area to be blocked. found,
* Coagulopathy, hepatic or renal failure,
* Allergic to a local anesthetic agent or one of the drugs used in the study,
* Having a history of chronic opioid and corticosteroid use,
* who cannot use the patient-controlled analgesia system and have a psychiatric disease,
* with operative time less than 20 minutes and more than 120 minutes for better standardization of studies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Postoperative opioid consumption | Postoperative 24 hours
  First 24 hours total morphine consumption with patient controlled analgesia

SECONDARY OUTCOMES:
Numerical Rating Scale | Postoperative 24 hours
  To determine the pain of the patients at rest and passive-active moving at the 1st, 3rd, 6th, 12th, 18th and 24th hours postoperatively with Numerical Rating Scale (NRS).The NRS is a segmented numerical version in which the respondent selects an integer (0-10) that best reflects the intensity of their pain. 0: no pain 1-3: mild pain 4-6: moderate pain 7-10: severe pain.
Timed up and go test (TUG) | at 24th hour
  TUG- evaluation of the time in seconds for the patient to get up from the chair and walk 3 meters and return to the chair again
Quadriceps muscle strength | at 24th hour
  will be evaluated in a scale between 1-5 (1:lowest; 5:normal)

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Süren, Professor, Study Chair — Samsun Research and Education Hospital
Locations (1):
- Samsun Research and Education Hospital, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Researched data and statistical analyzes will be available from the journal in which the clinical study was published

REFERENCES:
- [Result] Seo SS, Kim OG, Seo JH, Kim DH, Kim YG, Park BY. Comparison of the Effect of Continuous Femoral Nerve Block and Adductor Canal Block after Primary Total Knee Arthroplasty. Clin Orthop Surg. 2017 Sep;9(3):303-309. doi: 10.4055/cios.2017.9.3.303. Epub 2017 Aug 4. PMID 28861197
- [Result] Desmet M, Balocco AL, Van Belleghem V. Fascia iliaca compartment blocks: Different techniques and review of the literature. Best Pract Res Clin Anaesthesiol. 2019 Mar;33(1):57-66. doi: 10.1016/j.bpa.2019.03.004. Epub 2019 Apr 17. PMID 31272654
- [Result] Vermeylen K, Soetens F, Leunen I, Hadzic A, Van Boxtael S, Pomes J, Prats-Galino A, Van de Velde M, Neyrinck A, Sala-Blanch X. The effect of the volume of supra-inguinal injected solution on the spread of the injectate under the fascia iliaca: a preliminary study. J Anesth. 2018 Dec;32(6):908-913. doi: 10.1007/s00540-018-2558-9. Epub 2018 Sep 24. PMID 30250982
- [Result] Pehora C, Pearson AM, Kaushal A, Crawford MW, Johnston B. Dexamethasone as an adjuvant to peripheral nerve block. Cochrane Database Syst Rev. 2017 Nov 9;11(11):CD011770. doi: 10.1002/14651858.CD011770.pub2. PMID 29121400